CLINICAL TRIAL: NCT01174082
Title: Phase II Trial of ID-Specific Donor Vaccinated Lymphocyte Infusion for Patients With Myeloma Relapsing or Failing to Achieve a Complete Remission After an Allogenic Transplant
Brief Title: Trial of ID-Specific Donor Vaccinated Lymphocyte Infusion for Patients With Myeloma Relapsing or Failing to Achieve a Complete Remission After an Allogenic Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2004-0660; NCI-2012-01781 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Vaccine; Lymphocyte Infusion
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Blood Component Removal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- KLH Vaccine (Patient) (Experimental): After DLI on same day, patients receive vaccine according to donor randomization (the same type of vaccine that their donors received).
  Interventions: Biological: KLH Vaccine; Drug: GM-CSF; Procedure: Donor Lymphocyte Infusion (DLI)
- KLH-id Vaccine (Patient) (Experimental): After DLI on same day, patients receive vaccine according to donor randomization (the same type of vaccine that their donors received).
  Interventions: Biological: KLH-id Vaccine; Drug: GM-CSF; Procedure: Donor Lymphocyte Infusion (DLI)
- KLH Vaccine (Donor) (Experimental): Donor Group 1: (non-specific vaccination) vaccinated with KLH only vaccine 0.5 cc subcutaneously, 3 times on weeks -8, -6 and -2 prior to donor lymphocyte collection.
  Interventions: Biological: KLH Vaccine; Drug: GM-CSF; Procedure: Apheresis
- Vaccine KLH-id (Donor) (Experimental): Donor Group 2: (myeloma specific vaccination) vaccinated with KLH-id vaccine 0.5 cc subcutaneously, 3 times on weeks -8, -6 and -2 prior to donor lymphocyte collections.
  Interventions: Biological: KLH-id Vaccine; Drug: GM-CSF; Procedure: Apheresis

INTERVENTIONS:
Biological: KLH Vaccine — Donor: 0.5 cc subcutaneously, 3 times on weeks -8, -6 and -2 prior to lymphocyte collection.
  Patient: 0.5 cc subcutaneously, 3 times immediately after infusion of donor cells (DLI), and again 4 and 8 weeks post DLI.
  Arms: KLH Vaccine (Donor); KLH Vaccine (Patient)
Biological: KLH-id Vaccine — Donor: 0.5 cc subcutaneously, 3 times on weeks -8, -6 and -2 prior to donor lymphocyte collection.
  Patient: 0.5 cc subcutaneously, 3 times immediately after infusion of donor cells (DLI), and again 4 and 8 weeks post DLI.
  Arms: KLH-id Vaccine (Patient); Vaccine KLH-id (Donor)
Drug: GM-CSF — 250 mcg/m2 subcutaneously daily for 4 days after each vaccine
  Other Names: Sargramostim; Leukine
Procedure: Apheresis — Day 0 (day of lymphocyte collection) donors undergo a steady state pheresis to obtain lymphocytes.
  Arms: KLH Vaccine (Donor); Vaccine KLH-id (Donor)
Procedure: Donor Lymphocyte Infusion (DLI) — Day 0, infusion to patient of collected donor cells.
  Arms: KLH Vaccine (Patient); KLH-id Vaccine (Patient)

SUMMARY:
The goal of this clinical research study is to learn if vaccinating a donor with your purified myeloma protein and then injecting it back into you will help your immune system control the multiple myeloma.

DETAILED DESCRIPTION:
A vaccine will be made of tumor protein taken from your plasma (liquid part of the blood) and KLH (a protein designed to increase the immune response of the vaccine). By vaccinating your brother or sister with protein made from the tumor, researchers hope to increase the antitumor effect of the stem cells. KLH is used to help the immune response.

Study Treatment Schedule:

If you are found to be eligible to take part in this study, you and your brother or sister will receive a vaccine with KLH. This research involves various steps. In Step 1, a large sample of your plasma will be collected through a vein using a blood separator device. This plasma will be sent to the MD Anderson GMP lab to prepare the vaccine. It takes about 3 months to create your myeloma-specific vaccine. It takes about 3 months to prepare enough vaccine for the next phases of the study.

In Step 2, your brother or sister will receive the vaccine with KLH as an injection under the skin 8 weeks, 6 weeks, and 2 weeks before collection of his/her lymphocytes (immune fighting cells). After each injection, your brother or sister will receive an injection of a medication called GM-CSF that helps the body's response to the vaccine. GM-CSF is given under the skin near the site of the vaccination every day for 4 days, starting the day of the vaccination.

In Step 3, your brother or sister will have apheresis. During apheresis, their blood is passed through a "cell separator" and the lymphocytes (immune fighting cells) are collected. A portion of these cells will be given to you on this day. You will get these cells through a vein while the remainder is stored and frozen for research and/or use later on if you fail to respond to the first infusion.

In Step 4, you will receive the vaccine with KLH. It will be given under the skin immediately after you get the infusion of donor cells, and again 4 and 8 weeks after the lymphocyte infusion. After each vaccine, you will receive an injection of a medication called sargramostim (GM-CSF) that helps the body's response to the vaccine. GM-CSF is given under the skin near the site of the vaccination every day for 4 days, starting the day of the vaccination.

If after 6 months you are not responding to the vaccine, you will be allowed to receive 3 additional vaccines, as long as you did not develop graft versus host disease or any other serious side effects to the first vaccine. The vaccines and follow-up schedule is exactly like the first.

Study Visits:

Within 10 days before you receive the infusion of your donor's cells and within 72 hours before each vaccine injection, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs.
* You will be checked for possible reactions to your treatment, including graft-versus-host disease (GVHD). Infused donor cells may react against your body.
* You will be asked about any side effects you may have had since the first vaccine injection.
* Blood (about 6-12 teaspoons) will be drawn for routine tests and to check your kidney and liver function, as well as the status of your immune system. Part of the blood will be used to test for CMV, hepatitis B, hepatitis C, HIV, HTLV, syphilis, West Nile virus, sickle cell anemia, and Chagas disease. Part of the blood collection will also be used for a pregnancy test for females who are able to have children. To continue to receive infusions of your donor's cells, the pregnancy test must be negative.
* You will have x-rays or bone marrow aspirates and biopsies to assess the response of your disease.

These visits will require 1 day of your time.

Long-Term Follow-Up:

Once a month during Months 3, 6, 12, 18, and 24 months after your last vaccine, the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your vital signs.
* You will be checked for possible reactions to your treatment, including GVHD.
* Blood (about 6-12 teaspoons) will be drawn to check your kidney and liver, function as well as the status of your immune system. Part of the blood collection will also be used for a pregnancy test for females who are able to have children. To continue to receive infusions of your donor's cells, the pregnancy test must be negative.
* You will have a bone marrow biopsy and aspiration. It may be repeated more often, if your doctor thinks it is needed.

If you are not able to return to MD Anderson, your study doctor may agree to allow you to have these tests and procedures at your local doctor's office. Your local doctor will need to send the results to research staff at MD Anderson.

Once a year, starting 2 years after you receive the last infusion of your donor's cells, you will be contacted by phone to check on your health status.

Length of Study Participation:

You will be considered off study after 5 years. You will be taken off study at any time if lymphocytes cannot be collected, not enough lymphocytes can be collected, your doctor thinks it is needed, the recipient is not able to receive the vaccine, the study doctor thinks it is in your best interest, you need a treatment that is not allowed while on this study, you are unable to keep appointments, or you have intolerable side effects.

This is an investigational study. The myeloma-specific vaccine is not FDA approved or commercially available, and it has been authorized for use in research only. Up to 10 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient: Patient with IgG1, IgG2, or IgG4 Multiple Myeloma who has received or planning to receive an allogeneic progenitor cell transplant from a HLA compatible related donor (either 6/6 or 5/6 related donor).
2. Recipient: Have evidence of persistent or relapsing disease as demonstrated by persistent serum peak (by either standard protein electrophoresis, immune fixation or free light chain assays) or marrow infiltration. Serum peak must be greater or equal than 0.2 gm/dl and represent more than 70% of the specific immunoglobulin subtype. Patients who have adequate amount of monoclonal idiotype protein previously cryopreserved on prior departmental laboratory protocols are also eligible to be registered for vaccine production using the cryopreserved samples.
3. Recipient: Able to sign written informed consent.
4. Recipient: Age up to 70 years.
5. Recipient: Zubrod PS >/=2.
6. Recipient: Have no serious organ dysfunction as defined by serum creatinine <2.5 mg/dL, serum bilirubin <3 x upper limit of normal, SGPT <4 x upper limit of normal.
7. Recipient: Negative donor infectious disease panel: Hepatitis B surface antigen (HBsAg), Anti-Hepatitis B core antibody (HBcAb), Anti-Hepatitis C Virus antibody (HCV Ab), Anti-Human Immunodeficiency Virus (HIV) antibody (HIV 1/2 type O Ab), Anti-Human T cell lymphotrophic Virus (HTLV) antibody (HTLV I/II Ab), Rapid Plasma Reagen (RPR), Cytomegalovirus antibody (CMV), HCV/HIV Nucleic Acid Test, West Nile Virus Nucleic Acid Test, Sickledex, T Cruzi AB. Additional tests shall be performed as required to assess the possibility of transmission of other infectious or non-infectious diseases.
8. Recipient: Negative serum Beta HCG test in a women with child bearing potential (not post-menopausal for 12 months or no previous surgical sterilization) and willing to use an effective contraceptive measure while on study. Mothers should not breastfeed during the study.
9. Donor: Able to sign written informed consent and be willing to provide donor lymphocytes.
10. Donor: Age 18 - 75 years
11. Donor: No physical contraindications to lymphocyte collection (i.e. severe atherosclerosis, auto-immune disease, cerebrovascular accident, prior malignancy less than 5 years ago other than non-melanoma skin cancer treated with surgery). Donors with severe atherosclerosis by history will receive a cardiology consult and be judged eligible on a case by case basis.
12. Donor: Negative donor infectious disease panel: Hepatitis B surface antigen (HBsAg), Anti-Hepatitis B core antibody (HBcAb), Anti-Hepatitis C Virus antibody (HCV Ab), Anti-Human Immunodeficiency Virus (HIV) antibody (HIV 1/2 type O Ab), Anti-Human T cell lymphotrophic Virus (HTLV) antibody (HTLV I/II Ab), Rapid Plasma Reagen (RPR), Cytomegalovirus antibody (CMV), HCV/HIV Nucleic Acid test. Additional tests shall be performed as required to assess the possibility of transmission of other infectious or non-infectious diseases.
13. Donor: Negative serum Beta HCG test in a woman with child bearing potential (not post-menopausal for 12 months or no previous surgical sterilization) must use an effective method of contraception until at least 1 month after lymphocyte collection. Mothers should not breastfeed during the study.

Exclusion Criteria:

1) Recipient with IGg3 Multiple Myeloma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07-20 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffar H. Qazilbash, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Recipient: Vaccine + DLI
- Donor: Vaccine
Period: Overall Study
Arm/Group | Recipient | Donor
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recipient | Donor | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Partial Response(PR) and Complete Response(CR) in Patients Receiving DLI From an ID-specific Vaccinated Donor
Description: PR defined as 50% reduction disease including serum monoclonal paraprotein and CR defined as absence of original monoclonal paraprotein in serum and urine.
Time Frame: DLI up to 5 years post DLI
Population: The donor participant was to supply the cell product to manufacturer the vaccine. The donor has no disease and therefore cannot be analyzed for a response.
Measure: Count of Participants; unit: Participants
Arm/Group | Recipient | Donor
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years post start of treatment
Groups:
- Recipient: KLH vaccine + DLI
- Donor: KLH vaccine
Arm/Group | Recipient | Donor
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Recipient (N=1) | Donor (N=1)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Abd cramping (Gastrointestinal disorders) | 1 | 0
Insomnia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Decreased Platelet (Blood and lymphatic system disorders) | 1 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fever (General disorders) | 1 | 1
Chills (General disorders) | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hearing Loss (Ear and labyrinth disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Neuropathy (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT01174082/Prot_SAP_000.pdf